CLINICAL TRIAL: NCT01297816
Title: Evaluation of Minocycline Neuro Protective Role in Retinal Detachment Surgery
Brief Title: Evaluation of Neuroprotective Effect of Minocycline
Acronym: minocyclin &RD
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Responsible Party: Mohsen Azarmina, Ophthalmic Research center
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: 89122
Record Dates: First submitted 2011-01-19; First posted 2011-02-17 (Estimated); Last update posted 2011-02-17 (Estimated); Status verified 2010-12

CONDITIONS: Retinal Detachment
MeSH Terms: conditions — Retinal Detachment | interventions — Minocycline

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- placebo (Placebo Comparator): 100mg-
  Interventions: Drug: placebo
- minocyclin (Placebo Comparator)
  Interventions: Drug: Minocycline

INTERVENTIONS:
Drug: placebo — 100mg,BD, fo three month
  Arms: placebo
Drug: Minocycline — 100mg
  Arms: minocyclin

SUMMARY:
This process appears as a incredible and progressive event that will not stop till reattachment of RPE and neurosensory retina happened .

Process of degeneration begins from first hours of RD (Retinal Detachment) establishment Neuroprotection of photoreceptor following RD is a novel and debatable discussion encountered in recent years .

How to stop this phenomena and neuroprotective agent role in this issue are a new interest of researcher.

In the study the investigators are planning to perform a clinical trial to demonstrate the minocycline neuroprotective effect in a double blind design as this impact has been implicated previously in a animal study

ELIGIBILITY:
Inclusion Criteria:

* age over 8 years old
* gender of both sex
* normal liver and renal function
* informed consent received from all patients
* no pregnancy and no lactation
* minimal sun exposure

Exclusion Criteria:

* old RD
* diabetic retina
* previous retinal surgery CRF& liver disfunction RD + PVR > B Hyper sensitivity to tetracycline History previous MPC or PRP Patients unsuccessful SB (retina is off )

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2010-12; Primary Completion 2010-12 (Estimated); Study Completion 2011-04 (Estimated)

PRIMARY OUTCOMES:
BCVA | changes of BCVA in 3 month
  outcome method of measurement: Snellen chart

SECONDARY OUTCOMES:
finding of ERG changes | 3 months
  outcome method of measurement: ERG( testes)
finding of OCT changes | 3 months
  outcome method of measurement: OCT
finding of FAF changes | 3 months
  outcome method of measurement: FAF( testes)

CONTACTS AND LOCATIONS:
Locations (1):
- Labbafinejad medical center, Tehran, Tehran Province, Iran